CLINICAL TRIAL: NCT02634138
Title: Neuromuscular Electrical Stimulation in Patients With Critical Limb Ischaemia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Halted prematurely
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14HH2036
Record Dates: First submitted 2015-12-01; First posted 2015-12-17 (Estimated); Last update posted 2019-06-06 (Actual); Status verified 2019-06

CONDITIONS: Peripheral Arterial Disease; Critical Limb Ischaemia
Keywords: Peripheral Vascular Disease; Critical Limb Ischaemia
MeSH Terms: conditions — Peripheral Arterial Disease; Chronic Limb-Threatening Ischemia; Peripheral Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention (Experimental): Revitive IX Neuromuscular Electrical Stimulation Device
  Interventions: Device: Revitive IX

INTERVENTIONS:
Device: Revitive IX — A foot plate Neuromuscular Electrical Stimulation Device

SUMMARY:
This study will assess the benefit of a neuromuscular electrical stimulation device in patients suffering from symptoms and effects of critical limb ischaemia.

DETAILED DESCRIPTION:
The circulation of blood around the body is dependent on effective pumping of the heart. Patients with arterial insufficiency are known to have poor circulation in their lower legs and feet leading to various complications such as swelling and painful legs and reduced healing of injuries.

Peripheral arterial disease (PAD) can be defined as a narrowing of the arteries reducing blood flow. It is most commonly due to atherosclerosis, and has associations with heart disease, stroke, and diabetes. Its incidence is estimated at 7-14% in the general population, increasing with age to about 20% in the over-seventies. It is associated with effects on mobility, skin condition and quality of life. Symptoms include pain in the legs on walking (intermittent claudication), pain at rest (particularly at night), gangrene, and limb loss. Management of PAD is based on encouraging exercise, and modification of risk factors such as smoking, high blood pressure, high cholesterol and diabetes.

In patients with PAD, exercise tolerance is often limited. Severe symptoms and disease can be treated via such as balloon angioplasty, stenting or surgical bypass, but these procedures have risk. There also remains a percentage of patients who are not suitable for revascularisation, and have only a few options such as amputation available to them.

Some trials have shown that increasing the blood flow in the legs over time using medical devices (intermittent pneumatic compression, muscle stimulators), in addition to maximal medical and surgical therapy, can increase claudication distance, absolute walking distance, decrease rest pain, and reduce amputation rates. In the investigators unit it has become apparent that there are an increasing number of medical devices available for circulatory support, either as an inpatient, out-patient, or a member of the general public. The supporting evidence for these is variable in scientific and clinical content or relevance, and requires clinical trials to evaluate further.

Revitive activates the pumping action of leg muscles by providing electrical muscle stimulation to cause foot muscle contraction and relaxation which squeezes blood back towards the heart, improving circulation.

The investigators wish to evaluate whether NMES using this device has the same beneficial effects in patients with critical limb ischaemia.

ELIGIBILITY:
Inclusion Criteria:

* Willing, able, and committed to participate in the procedures for the full length of the study.
* All ethnic groups, male or female above the age of 18 years.
* Diagnosis of non-reconstructable arterial disease and critical limb ischaemia (with a minimum of duplex ultrasound and an MDT discussion to have reached this diagnosis)
* Be of non-childbearing potential; OR using adequate contraception and have a negative urine pregnancy test result within 24 hours if appropriate before using the study device.
* Blood pressure currently under moderate control (< 160/100mmHg)
* History of uncomplicated cardiovascular events beyond 3 months.
* No current foot ulceration

Exclusion Criteria:

Patients meeting any of the following criteria are to be excluded:

* Has an unstable condition (eg, psychiatric disorder, a recent history of substance abuse) or otherwise thought to be unreliable or incapable of complying with the study protocol.
* Has any metal implants
* Pregnant
* Has peripheral neuropathy
* Has a cardiac pacemaker or defibrillator device
* Has recent lower limb injury or lower back pain
* Has current foot ulceration or other skin ulcers
* Has foot deformities
* Has any disorder that, in the opinion of the Investigator, might interfere with the conduct of the study
* Ankle-Brachial Pressure Index >0.9

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-11; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Pain Score | 6 weeks
  Change in pain score with device use over a 6 week period. Measure by a visual analogue scale of pain with 0 = no pain and 10 = maximum pain

SECONDARY OUTCOMES:
Major amputation rate | 6 weeks
  Identify if and number of major amputations carried out during study period.
Flow rate in Femoral Artery | Day 1 then at 6 weeks
  Duplex ultrasound guided measurement of femoral artery flow rate whilst using the device on day 1 and then 6 weeks later during follow up visit.
Femoral artery diameter | Day 1 and at 6 weeks
  Duplex ultrasound guided measurement of femoral artery diameter whilst using the device on day 1 and then 6 weeks later during follow up visit.
Disease specific questionnaire - VascuQoL | Day 1 and at 6 weeks
  Change of disease specific Quality of Life (QoL) measure from baseline to 6 weeks.
Short Form - 36 (SF-36) | Day 1 and at 6 weeks
  Change ofSF-36 Quality of Life (QoL) score from Day 1 to 6 weeks.
EuroQol - EQ5D | Day 1 and at 6 weeks
  Change of EQ5D Quality of Life (QoL) score from Day 1 to 6 weeks.
Patient compliance using diary of device use | 6 weeks
  Check the frequency of device use over the 6 week study period.

CONTACTS AND LOCATIONS:
Overall Officials: Alun H Davies, BA BMChB MA, Study Chair — Imperial College London
Locations (1):
- Imperial College London - Charing Cross Hospital, London, United Kingdom